CLINICAL TRIAL: NCT03305991
Title: The Role of Maternal TB Infection for Adverse Pregnancy and Infant Health Outcomes in Ethiopia - a Long-term Prospective Cohort Study
Brief Title: Tuberculosis Infection in Women of Reproductive Age and Their Infants
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Per Bjorkman, Professor, Lund University
Other Study IDs: LundU-2015
Record Dates: First submitted 2017-10-02; First posted 2017-10-10 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Tuberculosis; Pregnancy Complications
Keywords: tuberculosis; pregnancy; ethiopia
MeSH Terms: conditions — Tuberculosis; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen aliquots of plasma samples stored at Adama Regional Laboratory, Ethiopia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Women living in low-income countries are at elevated risk of death in connection to pregnancy, as well as infants born to women in such settings. It is probable that several factors are involved, such as poverty, lack of education and access to healthcare. Infectious diseases constitute important threats to maternal health in resource-limited settings. Tuberculosis (TB) is reported to be the third leading cause of maternal death globally. Furthermore, TB can be transmitted from mother to child during pregnancy, with high risk of severe consequences for the infant. Despite these data, neither the role of TB in relation to co-existing risk factors for adverse pregnancy outcomes, nor the mechanisms involved, are well understood. It is likely that TB interacts with other characteristics, in particular socio-economic condition and HIV infection, which could obscure associations between TB and pregnancy outcomes. For this reason, it is critical to design studies so that the independent role of TB can be deduced.

This project aims to investigate how TB infection in women affects the risk of adverse pregnancy outcomes in relation to co-existing factors, and how exposure to TB infection may impact growth and development of infants born to women with TB. In addition, mechanisms in which TB and the immune system during pregnancy will be explored.

The project is conducted at public health facilities in Ethiopia, where 2 000 women have been recruited during antenatal care. These women will be followed until 5 years after delivery, along with their offspring born during the study period. Detailed data is collected at inclusion and at study visits during follow-up, with submission of samples for TB testing and immunological analyses.

Better knowledge on the characteristics of TB infection in association with pregnancy, and how TB affects maternal and child health, can be used to construct new guidelines for management of TB in women of fertile age. This may contribute to reductions in adverse pregnancy outcomes, including maternal and infant deaths.

DETAILED DESCRIPTION:
Objective The overall objective of this project is to investigate longitudinal patterns and consequences of tuberculosis (TB) infection in a prospective cohort of women recruited during pregnancy. The relation between maternal TB infection and pregnancy outcomes, as well as infant health and development, will be evaluated over time.

Specific aims

1. To determine whether maternal TB infection is associated with adverse pregnancy outcomes
2. To determine the excess risk of incident active TB during pregnancy and post-partum, with regard to the prevalence of latent TB infection at registration in antenatal care
3. To investigate long-term health and survival in infants in relation to maternal TB and adverse pregnancy outcomes

Methods Study setting and participants This project is conducted in public health facilities in the city of Adama, Central Ethiopia. Participants are recruited and followed at antenatal care (ANC) clinics until delivery. After delivery their children are followed at clinics for extended program for immunization (EPI); continued follow-up of the mothers after the first post-natal visit also takes place in these clinics.

All study procedures, including interviews, physical examination, and collection of informed consent, are performed by health facility staff (nurses and midwives) in the respective clinics. Biological samples including blood and sputum are collected at the respective health facility laboratory. Study samples are transported to the Adama Regional Laboratory. At this laboratory, additional analyses and storage of plasma will be done.

For supervision and monitoring of data collection, as well as for data entry, the project uses staff and infrastructure in a field research station which has been established in Adama since 2010 by the research group.

Study procedure Both scheduled and unscheduled study visits can occur for participants in this project. Scheduled study visits coincide with routine antenatal and postnatal visits and visits at the EPI clinics for the infant's immunization following National guidelines. Unscheduled visits occur in case of symptoms suggestive of active TB (according to the study definitions) in the pregnant/postnatal/non-pregnant woman, or in the child, at any time in between these routine visits.

Antenatal care visits At inclusion, structured information on socio-demographic conditions, education, occupation, and poverty indicators is collected; as well as medical history (in particular for obstetric, gynecological and TB-related details). Physical and obstetric examination is performed. Apart from the study procedures and investigations, participants will receive care according to current Ethiopian ANC guidelines.

At the inclusion visit blood samples are obtained for routine care and for study specific investigations from all participants. At the health facility laboratory, the following analyses are performed: HIV rapid test, urine dipstick. Ten mL of venous blood is collected. This sample is used for analysis of complete blood count, blood/Rh group, syphilis serology, creatinine and fasting glucose. The remaining plasma is aliquoted and stored at -80° C for research analyses that are performed at the completion of inclusion. Blood is collected separately for QuantiFERON TB Plus (QFT) testing, in order to determine the prevalence of LTBI. For the last 500 women included in the study, QFT testing is repeated at the 3rd antenatal care visit. From HIV positive women blood for viral load and CD4 count is drawn at each scheduled visit pre- and post-delivery except from 2nd and 3rd antenatal care visit.

Participants are followed up four times in accordance with WHO recommended focused antenatal visits until delivery or term of pregnancy. They are also instructed to contact the study clinic in between these visits in case of health-related events. In case of delivery (or other unintended termination of pregnancy) in another place than any of the study health facilities, they are asked to communicate this to their study site for further follow-up examinations.

All participants with suspected active TB according to the study definition (irrespective of Quantiferon results) at enrolment and/or during follow up are asked to submit samples for bacteriological TB investigations. These encompass liquid culture, smear microscopy and PCR (using Xpert MTB/RIF technique). All these tests are performed on two consecutive morning sputum samples. Moreover, acquisition of blood for QuantiFERON testing is repeated for all women investigated for suspected active TB.

Stored aliquots of Mtb-incubated plasma will be analyzed at the end of inclusion for potential blood biomarkers of TB infection during pregnancy. These analyses will be performed using ELISA and/or Luminex technique, and they will include the following markers of immune activation and inflammation: C-reactive protein (CRP), neopterin, soluble urokinase-plasminogen activator receptor (suPAR), interferon-inducible protein 10 (IP-10).

Postpartum follow-up visits for women Further follow-up visits for women are scheduled for 6 weeks and 9 months after delivery or termination of pregnancy, coinciding with the routine child visits for immunization. The first postnatal visit takes place at the ANC clinic, whereas all subsequent visits take place at the respective EPI clinics (where infant follow-up also occurs). At the 6 week postnatal visit details on delivery outcome are recorded.

For investigation of long-term health effects after delivery, participants will be asked to come for further annual visits with similar assessments until 54 months after termination of pregnancy. At all follow-up visits symptoms and signs on physical examination will be recorded using structured questionnaires.

At inclusion, and repeatedly on scheduled follow-up visits, participants are informed about symptoms and signs that may indicate active TB. Study subjects are instructed to contact the study site clinic (ANC during antenatal period, EPI during postnatal period) directly if they develop such symptoms for unscheduled study visits (in order to assess incident active TB during follow-up).

At all visits, whether scheduled or unscheduled, bacteriological testing (smear microscopy, Xpert MTB/RIF assay, and liquid culture) is performed according to the study protocol in case study criteria for suspected active TB are met. These tests are performed on two morning sputum samples.

In case study participants do not come for their scheduled study visits they are contacted by phone by the study site staff and/or the research study team. If the participant cannot be reached, her contact person is contacted by phone. At mid-time in between the scheduled visits, women are contacted by phone by a member of the local research team to assess whether any health events or symptoms compatible with TB have occurred.

Repeated sampling for QFT testing will be performed for all women at 4 years after inclusion (irrespective of previous QFT results), with storage of incubated plasma for further analysis of immune markers of TB infection.

Follow-up visits for infants If consent has been provided by the mother, infants are registered and included in a separate infant follow-up cohort as soon as possible after birth. Birth details, including delivery method, weight, length, APGAR score, and head circumference are registered at inclusion of the infant. Follow-up of included infants takes place in the EPI clinic at the respective study health facilities. Follow-up visits are scheduled at the same time interval as the mother, i.e. at 6 weeks and 9 months and subsequently at annual intervals congruent with the mothers until four and a half year after birth. The two first visits coincide with routine immunization visits. On all study visits, parameters of growth, nutritional and neurological development are recorded using structured questionnaires. In addition, data on socio-demographic characteristics, health-related events and feeding details are recorded, as well as data on known or suspected exposure to TB.

At inclusion, and repeatedly on scheduled follow-up visits, caretakers are informed about symptoms and signs that may indicate active pediatric TB. Study infant caretakers are instructed to contact the study site EPI clinic directly if the infants develop such symptoms for unscheduled study visits (in order to assess incident active TB during follow-up).

If criteria for suspected TB are met at any time during follow-up bacteriological investigations (liquid culture, PCR and microscopy) will be performed on gastric lavage specimens (or cerebrospinal fluid in case of suspected meningitis; or fine-needle lymph node aspirates in case of peripheral lymphadenopathy). These investigations will be performed by trained health care staff at the Department of Pediatrics, Adama Regional Hospital.

Stored aliquots of plasma will be analyzed at the end of inclusion for potential blood biomarkers of TB in young children. These analyses will be performed using ELISA and Luminex technique, and they will include the following markers of immune activation and inflammation: C-reactive protein (CRP), neopterin, soluble urokinase-plasminogen activator receptor (suPAR).

In case infant participants do not come for their scheduled study visits their caretakers are contacted by phone by the study site staff and/or the research study team. If the caretaker cannot be reached, the contact person is contacted by phone. At mid-time in between the scheduled visits, caretakers are contacted by phone from a study investigator to assess whether any health events or symptoms compatible with TB have occurred in the infant.

Study definitions Suspected adult active TB is defined as any of the following symptoms or findings: Cough, fever, night sweating, weight loss (except following delivery), chest pain, reduced Karnofsky performance score (after pregnancy), peripheral lymph node enlargement, abdominal distension and/or abdominal mass (during study periods without pregnancy).

Suspected pediatric active TB is defined as any of the following symptoms or findings: Cough, fever, night sweating, chest pain, peripheral lymph node enlargement, abdominal distension and/or mass, weight loss, poor growth development, failure to thrive, acute or chronic malnutrition, neck stiffness, seizures, and loss of consciousness Latent TB infection is defined as a positive QuantiFERON® TB Gold Plus result (according to the manufacturer's reference range), in the absence of confirmed active TB and/or national TB guideline criteria for clinically diagnosed TB.

Confirmed active TB is defined as any subject with a positive bacteriological result (as per the national TB guideline), irrespective of clinical manifestations.

Clinically diagnosed active TB is defined as any subject without positive bacteriological results for TB, but who fulfils national TB guideline criteria for clinically diagnosed TB, and who are referred for anti-TB treatment.

Adverse pregnancy outcomes are defined as maternal or infant death following inclusion until 3 months after unintended termination of pregnancy; preterm birth (before 37 gestational weeks); spontaneous abortion; PE (as defined by the International Society for the Study of Hypertension in Pregnancy; 25); IUGR; peri-partum hemorrhage.

Intra uterine growth restriction is defined as growth deviation of weight below 2 SD (-22% or below 3rd quartile) at birth.

Post-partum TB is defined as confirmed or clinically diagnosed active TB within the 6 months period following termination of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending antenatal care at any of the study facilities
* First antenatal care visit for current pregnancy
* Written informed consent
* Accepts HIV testing
* Residence in uptake area during pregnancy period

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women are eligible for inclusion
Study Population: Participants are identified at antenatal care clinics at three public health facilities. The study population consists of women of reproductive age who are identified and recruited in antenatal care and followed until delivery and 4 years post-partum. Children born to participants of the study are followed for 4 years after birth for assessment of survival, growth and development.
Sampling Method: Probability Sample
Enrollment: 2120 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse pregnancy outcomes | 2015-2023
  Reports of pregnancy outcomes of participating women, collected and assessed during study follow-up and categorized with regard to normal or adverse pregnancy outcomes

SECONDARY OUTCOMES:
Incidence of active tuberculosis in participants during pregnancy, post-partum period and periods outside pregnancy, respectively | 2015-2023
  Bacteriologically and/or clinically diagnosed cases of active tuberculosis during study follow-up, categorized with regard to timing in relation to pregnancy
Pattern of child growth with regard to maternal tuberculosis infection status during pregnancy | 2016-2023
  Growth curves of children born to participating women, recorded during study follow-up until 4 years of age
Incidence of tuberculosis infection in Ethiopian infants during the first four years of life | 2021-2023
  Latent and active tuberculosis at 4 years of age among children born to women in the study cohort

CONTACTS AND LOCATIONS:
Overall Officials: Per Bjorkman, MD, PhD, Principal Investigator — Lund University
Locations (3):
- Ethiopia (3):
  - Adama Health Center, Ādama
  - Adama Regional Hospital, Ādama
  - Gheda Health Center, Ādama

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Getahun H, Sculier D, Sismanidis C, Grzemska M, Raviglione M. Prevention, diagnosis, and treatment of tuberculosis in children and mothers: evidence for action for maternal, neonatal, and child health services. J Infect Dis. 2012 May 15;205 Suppl 2:S216-27. doi: 10.1093/infdis/jis009. Epub 2012 Mar 22. PMID 22448018
- [Background] Grange J, Adhikari M, Ahmed Y, Mwaba P, Dheda K, Hoelscher M, Zumla A. Tuberculosis in association with HIV/AIDS emerges as a major nonobstetric cause of maternal mortality in Sub-Saharan Africa. Int J Gynaecol Obstet. 2010 Mar;108(3):181-3. doi: 10.1016/j.ijgo.2009.12.005. Epub 2010 Jan 13. PMID 20070964
- [Background] Jana N, Vasishta K, Saha SC, Ghosh K. Obstetrical outcomes among women with extrapulmonary tuberculosis. N Engl J Med. 1999 Aug 26;341(9):645-9. doi: 10.1056/NEJM199908263410903. PMID 10460815
- [Background] Mathad JS, Bhosale R, Sangar V, Mave V, Gupte N, Kanade S, Nangude A, Chopade K, Suryavanshi N, Deshpande P, Kulkarni V, Glesby MJ, Fitzgerald D, Bharadwaj R, Sambarey P, Gupta A. Pregnancy differentially impacts performance of latent tuberculosis diagnostics in a high-burden setting. PLoS One. 2014 Mar 21;9(3):e92308. doi: 10.1371/journal.pone.0092308. eCollection 2014. PMID 24658103
- [Background] Kothari A, Mahadevan N, Girling J. Tuberculosis and pregnancy--Results of a study in a high prevalence area in London. Eur J Obstet Gynecol Reprod Biol. 2006 May 1;126(1):48-55. doi: 10.1016/j.ejogrb.2005.07.025. Epub 2005 Sep 9. PMID 16154251
- [Background] Rustveld LO, Kelsey SF, Sharma R. Association between maternal infections and preeclampsia: a systematic review of epidemiologic studies. Matern Child Health J. 2008 Mar;12(2):223-42. doi: 10.1007/s10995-007-0224-1. Epub 2007 Jun 19. PMID 17577649
- [Background] Rowe JH, Ertelt JM, Way SS. Foxp3(+) regulatory T cells, immune stimulation and host defence against infection. Immunology. 2012 May;136(1):1-10. doi: 10.1111/j.1365-2567.2011.03551.x. PMID 22211994
- [Background] Espinal MA, Reingold AL, Lavandera M. Effect of pregnancy on the risk of developing active tuberculosis. J Infect Dis. 1996 Feb;173(2):488-91. doi: 10.1093/infdis/173.2.488. PMID 8568319
- [Background] Whittaker E, Kampmann B. Perinatal tuberculosis: new challenges in the diagnosis and treatment of tuberculosis in infants and the newborn. Early Hum Dev. 2008 Dec;84(12):795-9. doi: 10.1016/j.earlhumdev.2008.09.005. Epub 2008 Sep 27. PMID 18823726
- [Background] Bekker A, Du Preez K, Schaaf HS, Cotton MF, Hesseling AC. High tuberculosis exposure among neonates in a high tuberculosis and human immunodeficiency virus burden setting. Int J Tuberc Lung Dis. 2012 Aug;16(8):1040-6. doi: 10.5588/ijtld.11.0821. Epub 2012 Jun 12. PMID 22691968